CLINICAL TRIAL: NCT02241642
Title: Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER II Study
Brief Title: Safety and Performance Study of Large Hole Vascular Closure Device
Acronym: FRONTIER-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P190-00; CIV-13-11-011700 (Other: BfArM - German Competent Authority)
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Percutaneous Common Femoral Artery Arteriotomy Closure
Keywords: Percutaneous vascular closure device; vascular closure device; Large hole closure device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): VIVASURE CLOSURE DEVICE™
  Interventions: Device: VIVASURE CLOSURE DEVICE™

INTERVENTIONS:
Device: VIVASURE CLOSURE DEVICE™ — Large hole vascular closure device

SUMMARY:
The purpose of this Clinical Investigation is to validate that the clinical use of the VIVASURE CLOSURE DEVICE™ is safe for the operator, patient and third parties, and to confirm its performance to percutaneously close femoral arterial puncture sites in the range of 18-24 F, post endovascular procedures.

This is a non-inferiority study based on safety. Safety will be assessed by incidence and severity of major complication rates directly related to the VIVASURE CLOSURE DEVICE™ up to 3 months from implantation is no worse than those associated with cut-down and sutured close.

DETAILED DESCRIPTION:
This study will be a prospective, multi-centred, non-randomized study to investigate the safety and performance of the VIVASURE CLOSURE DEVICE™. The study shall not be blinded prior to, during or post the procedure. All patients undergoing a procedure requiring an arteriotomy in the range of 18 to 24 F, via the common femoral artery will be screened against the inclusion/exclusion criteria. If the patient meets the requirements of the clinical investigation, they shall be invited to participate, provide informed consent and shall subsequently be assigned a subject number.

All subjects shall have an immediately post procedure, 24 hour, 1, 3 and 12 month follow-up assessment. Safety data from the follow-ups will be assessed by the Data Safety Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Each patient, or his or her guardian or legal representative, is willing to give informed consent
* Clinically indicated for an endovascular procedure involving access through the femoral artery, with an access puncture of 18 - 24 French (F)
* Females who are not pregnant or lactating, and not planning to become pregnant in ≤ 12 months

Exclusion Criteria:

* Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than one year
* Evidence of systemic bacterial or cutaneous infection
* Evidence of MRSA (Methicillin-resistant Staphylococcus aureus) and/or VRE (vancomycin-resistant Enterococci) colonisation
* Arterial access other than the common femoral artery
* Patients suffering with definitive or potential coagulopathy or platelet count less than 100,000/μl
* Patient with a haematocrit of less than 32 %
* A measured activated clotting time (ACT) of greater than 350 seconds immediately prior to sheath removal
* If patients are expected to be continuously treated with anticoagulation therapy post-procedure such that their ACT reading is expected to be elevated above 350 seconds for more than 24 hours after the procedure
* Evidence of arterial diameter stenosis greater than 20 % within 20 mm of the arteriotomy
* Circumferential calcification within 20 mm of the arteriotomy
* Use of systemic thrombolytic agents within 24 hours prior to or during the catheterisation procedure which cause the concentration of fibrinogen to be less than 100 mg/dl
* Patients in which the arteriotomy is less than 18 F or greater than 24 F
* Known allergy to any of the materials used in the device
* Currently enrolled in any other investigational clinical study, whereby the primary endpoint has not yet been achieved
* Patients judged unsuitable for surgical repair of the access site
* If puncture site is via a vascular graft
* If there is any indication that the puncture has been made in the profunda femoris or located less than 10 mm above the profunda femoris
* Patients with a common femoral artery lumen diameter of less than 7 mm
* Patients that have a lower extremity amputation from the ipsilateral or contralateral limb
* Patients that have undergone a percutaneous procedure using a non-absorbable vascular closure device (excluding suture mediated) for haemostasis in the ipsilateral leg
* Patients that have undergone a percutaneous procedure greater than 8 F in the ipsilateral leg, within the previous 90 days
* Patients that have undergone a percutaneous procedure of 8 F or less using an absorbable intravascular closure device for haemostasis, in the ipsilateral leg, within the previous 90 days
* Patients that have undergone a percutaneous procedure of 8 F or less using a suture mediated closure device for haemostasis, in the ipsilateral leg, within the previous 30 days
* Patients that have undergone a percutaneous procedure of 8 F or less using manual/mechanical pressure for haemostasis in the ipsilateral leg, within the previous 30 days
* Patients with an acute haematoma of any size, arteriovenous fistula or Pseudoaneurysm at the access site
* Significant blood loss/transfusion during interventional procedure or within 20 days of procedure requiring transfusion of greater than 4 units of blood
* Angiographic evidence of arterial laceration, dissection or stenosis within the external iliac or femoral artery before the use of the VCD
* Severe claudication, stenosis of the iliac artery > 50% or previous bypass surgery/stent placement in the region of the vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 3 months
  Incidence and severity of major complication rates (as defined by VARC-2) directly related to the VIVASURE CLOSURE DEVICE™ up to 3 months from implantation, is no worse than those associated with cut-down and sutured close

SECONDARY OUTCOMES:
Secondary Endpoint | 3 Months
  Incidence of minor complications (as defined by VARC-2) directly related to the VIVASURE CLOSURE DEVICE™ up to 3 months from implantation.

OTHER OUTCOMES:
Performance | Immediate
  Technical success rate for the VIVASURE CLOSURE DEVICE™

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med Giovanni Torsello, MD, Principal Investigator — St Fraziskus Hospital, Muenster, Germany
Locations (9):
- University Hospital Antwerp (UZA), Edegem, Belgium
- Germany (5):
  - The Charité - Universitätsmedizin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Leipzig, Leipzig
  - St Franziskus Hospital, Münster
- Ireland (2):
  - Blackrock Clinic, Blackrock
  - St James Hospital, Dublin
- St George's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No